CLINICAL TRIAL: NCT04495166
Title: Smartphone-Assisted Brief Behavioral Intervention for Pregnant Women With Depression
Brief Title: A Smartphone-Assisted Brief Behavioral Intervention for Pregnant Women With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Grand Challenges Canada (Other); Fundação Maria Cecilia Souto Vidigal (Other)
Responsible Party: Principal Investigator, Guilherme Vanoni Polanczyk, MD PhD, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Motherly1; SB-POC-1810-20573 (Other Grant/Funding Number: Grand Challenge Canada)
Record Dates: First submitted 2020-07-23; First posted 2020-07-31 (Actual); Results first posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-11

CONDITIONS: Perinatal Depression
MeSH Terms: interventions — Psychotherapy, Brief

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motherly app with brief psychotherapy (Experimental): Participants in this arm will receive intervention via Motherly 1.0, an app that delivers behavioral activation strategies and psychoeducational content to promote changes in sleep, nutrition, and physical activity habits. It has also functionalities that help participants to engage in prenatal care, breastfeeding, and social support, and to stimulate child development. In addition will undergo brief Cognitive-Behavioral Therapy (CBT) with a focus on behavioral activation.
  Interventions: Behavioral: Motherly 1.0; Behavioral: Brief Psychotherapy
- Educational app (Active control) (Active Comparator): Participants in this arm will have access to a psychoeducational app (active control) which delivers content about gestation, maternal health and mental health, and child development. In addition, they will undergo will undergo brief Cognitive-Behavioral Therapy (CBT) with a focus on behavioral activation.
  Interventions: Behavioral: Brief Psychotherapy; Behavioral: Educational app

INTERVENTIONS:
Behavioral: Motherly 1.0 — A mobile app designed to promote life habits that have been shown to improve physical and mental health in pregnant women. The app consists of a package of specific and customized interventions defined by eight different modules: 1) Mental Health; 2) Sleep; 3) Nutrition; 4) Physical activity; 5) Social support; 6) Prenatal support; 7) Postnatal support, and 8) Library of pre and postnatal content. The app relies on extensive psychoeducational content delivered as tutorials, brief messages, and available as a library that can be read at the users' discretion; behavior monitoring using schedules, checklists, and notifications to help participants keep track of their health care visits, and schedule behavior activation activities; and gaming elements such as changes in background appearance to reflect participant's mood assessment and ratings of activities, and graphical and easy-to-use questionnaires for obtaining information (mood, nutrition habits).
  Arms: Motherly app with brief psychotherapy
Behavioral: Brief Psychotherapy — Brief Cognitive-Behavioral Therapy (CBT) with a focus on behavioral activation (BA). Participants will be guided by psychotherapists to plan, schedule, and engage in positively reinforcing activities, and will be aided to develop problem-solving strategies for circumventing barriers to completing scheduled activities. Implementation of these techniques will be conducted with the aid of the Motherly 1.0 for participants in the experimental arm; for participants in the control arm, BA will be implemented without the aid of Motherly 1.0. Throughout the four sessions, psychotherapists will monitor participants' adherence, answering questions about the strategies and providing support for solving problems or CBT techniques, such as cognitive restructuring, relaxation techniques, sleep hygiene, stress and anxiety management, among other evidence-based techniques might be used if appropriate to the case.
Behavioral: Educational app — A simplified version of the Motherly 1.0 app consisting of psychoeducational content about various aspects of pregnancy, maternal physical and mental health, and child development. Active intervention functionalities, such as behavioral activation, activity scheduling, sleep hygiene, among others, are NOT present in this simplified version of the app.
  Arms: Educational app (Active control)

SUMMARY:
Investigators developed Motherly 1.0, a smartphone app designed to treat and promote maternal mental health. A 2-arm parallel-randomized controlled clinical trial (RCT) will be conducted to test the efficacy of Motherly in conjunction with brief cognitive-behavioral therapy. 70 pregnant women between 16-40 years old will be recruited. Since all interventions will be conducted online, participants will be recruited from any Brazilian state or municipality. Participants will be randomly assigned to either receive intervention via app consisting of behavioral activation and psychoeducation to promote changes in sleep, nutrition, and physical activity habits, as well as to engage in prenatal care, breastfeeding, and social support, and to stimulate child development, in addition to brief cognitive-behavioral therapy (CBT) (n=35); or to a comparison group receiving an psychoeducational app (active control) with psychoeducational content about gestation, maternal health and mental health, and child development in addition to brief CBT (n=35). Duration of treatment will be eight weeks, during which participants in both groups will be assessed at the beginning (baseline; T0), weeks 3-4 (midpoint; T1), and week 8 (endpoint; T2) in order to evaluate treatment effects. A follow-up postnatal assessment will also be conducted when the child is three months of age (T3).

ELIGIBILITY:
Inclusion Criteria:

* women aged between 16-40 years;
* having a score of >7 on the Edinburgh Postnatal Depression Scale (EPDS);
* gestational age between 17-26 weeks;
* being literate;
* owning a functional smartphone with Android for personal use.

Exclusion Criteria:

* pregnancies classified as being at risk, fetal malformation, or congenital disease;
* visual, auditory or intellectual disabilities, or chronic diseases associated with fetal development alterations;
* severe and/or chronic mental disorder (e.g., schizophrenia, bipolar disorder, etc).

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 81 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2021-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Fatori, PhD, Principal Investigator — Medical School, University of Sao Paulo
Locations (1):
- Daniel Fatori, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sockol LE, Epperson CN, Barber JP. A meta-analysis of treatments for perinatal depression. Clin Psychol Rev. 2011 Jul;31(5):839-49. doi: 10.1016/j.cpr.2011.03.009. Epub 2011 Mar 27. PMID 21545782
- [Background] Graham JW, Olchowski AE, Gilreath TD. How many imputations are really needed? Some practical clarifications of multiple imputation theory. Prev Sci. 2007 Sep;8(3):206-13. doi: 10.1007/s11121-007-0070-9. Epub 2007 Jun 5. PMID 17549635
- [Derived] Zuccolo PF, Xavier MO, Matijasevich A, Polanczyk G, Fatori D. A smartphone-assisted brief online cognitive-behavioral intervention for pregnant women with depression: a study protocol of a randomized controlled trial. Trials. 2021 Mar 23;22(1):227. doi: 10.1186/s13063-021-05179-8. PMID 33757591

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via social media advertisements from August to September 2020. After demonstrating interest in the study, potential participants were referred to a website page where they were informed of the study's aims, procedures, assessments, and nature of the interventions. They responded to an online survey assessing eligibility criteria. Eligible participants were invited to a baseline assessment conducted via internet or telephone.
Pre-assignment Details: Three hundred and twenty (320) women registered online, but 188 did not meet eligibility criteria and one had a duplicated registration. Thirty-six (36) women were excluded in a brief telephone because they did not meet eligibility criteria or declined to participate in the study. Ninety-five (95) women were scheduled for baseline assessment, but 14 cancelled or missed the appointment. Eighty one (81) participants were enrolled and randomized to intervention (N=37) or active control (N=44).
Groups:
- Motherly App With Brief Psychotherapy: Participants in this arm received intervention via Motherly 1.0, an app that delivers behavioral activation strategies and psychoeducational content to promote changes in sleep, nutrition, and physical activity habits. It has also functionalities that help participants to engage in prenatal care, breastfeeding, and social support, and to stimulate child development. In addition, they underwent a brief Cognitive-Behavioral Therapy (CBT) protocol with a focus on behavioral activation.
- Educational App (Active Control): Participants in this arm had access to a psychoeducational app (active control) which delivers content about gestation, maternal health and mental health, and child development. In addition, they underwent a brief Cognitive-Behavioral Therapy (CBT) protocol with a focus on behavioral activation.
Period: Overall Study
Arm/Group | Motherly App With Brief Psychotherapy | Educational App (Active Control)
Started | 37 | 44
Completed | 30 | 41
Not Completed | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Motherly App With Brief Psychotherapy: Participants in this arm received intervention via Motherly 1.0, an app that delivers behavioral activation strategies and psychoeducational content to promote changes in sleep, nutrition, and physical activity habits. It has also functionalities that help participants to engage in prenatal care, breastfeeding, and social support, and to stimulate child development. In addition they underwent a brief Cognitive-Behavioral Therapy (CBT) protocol with a focus on behavioral activation.
- Total: Total of all reporting groups
Arm/Group | Motherly App With Brief Psychotherapy | Educational App (Active Control) | Total
Number analyzed (Participants) | 37 | 44 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (4.6) | 32.3 (4.9) | 32.5 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 44 | 81
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 25 | 26 | 51
  Non-white | 12 | 18 | 30
Number of people in the house [Mean (Standard Deviation); unit: people in the house] | 3.0 (1.2) | 2.8 (1.2) | 2.9 (1.2)
Participant has college degree or higher [Count of Participants; unit: Participants] | 22 | 30 | 52
Participant is working for pay [Count of Participants; unit: Participants] | 23 | 30 | 53
Family income in Brazilian Real [Mean (Standard Deviation); unit: Brazilian Reais (R$)] | 5108.8 (4434.7) | 4214.8 (3179.3) | 4623.1 (3805.8)
Participant is studying [Count of Participants; unit: Participants] | 12 | 16 | 28
Participant is married or in a stable relationship [Count of Participants; unit: Participants] | 33 | 38 | 71
Number of prenatal visits [Mean (Standard Deviation); unit: prenatal visits] | 3.8 (1.6) | 4.6 (1.8) | 4.3 (1.7)
Gestational age in weeks [Mean (Standard Deviation); unit: weeks] | 18.7 (2.8) | 19.9 (3.3) | 19.4 (3.1)
Participant diagnosed with high-risk pregnancy [Count of Participants; unit: Participants] | 13 | 7 | 20
Participant is receiving mental health treatment [Count of Participants; unit: Participants] | 10 | 8 | 18
Participant used alcohol during gestation [Count of Participants; unit: Participants] | 7 | 3 | 10
Participant used tobacco during gestation [Count of Participants; unit: Participants] | 3 | 3 | 6
Participant used cannabis during gestation [Count of Participants; unit: Participants] | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Maternal Prenatal Depression at Baseline, Midpoint, and Posttreatment (8 Weeks)
Description: Participants were assessed with the Edinburgh Postnatal Depression Scale (EPDS) at baseline, at 4 weeks, and at 8 weeks (posttreatment). (EPDS max-min scores=0-30, higher scores=worse outcome).
Time Frame: Baseline (T0), Weeks 3-4 (Midpoint, T1), Week 8 (Posttreatment, T2).
Population: In order to include participants that were not assessed in post-baseline assessments we used multiple imputation by chained equations (MICE) with 100 imputations (Graham et al., 2007). MICE models included information from all outcomes at T1, T2, and T3, as well as key baseline characteristics.
Measure: Mean (95% Confidence Interval); unit: score on EPDS
Arm/Group | Motherly App With Brief Psychotherapy | Educational App (Active Control)
Number analyzed (Participants) | 37 | 44
score on EPDS
  T0 | 17.3 [15.8 to 18.8] | 16.8 [15.5 to 18.1]
  T1 | 12.5 [10.8 to 14.2] | 12.1 [10.5 to 13.6]
  T2 | 11.1 [9.3 to 13.0] | 10.8 [9.1 to 12.4]
Statistical Analysis 1: Comparison: Motherly App With Brief Psychotherapy vs Educational App (Active Control); The sample size was calculated based on an effect size of 0.65 on depression, which is based on a previous meta-analysis (Sockol et al., 2011). Sample size calculation considered a difference in means between two independent groups, probability of type I error of 5%, statistical power of 80%, a two-tailed test, and a dropout rate of 15%; Test type: Superiority; p = 0.757, t-test, 2 sided — Statistical tests were 2-sided and p values <0.05 were considered statistically significant; To include participants that were not assessed in post-baseline assessments we used multiple imputation by chained equations with 100 imputations

2. Secondary Outcome: Change in Maternal Prenatal Anxiety From Baseline to Posttreatment (8 Weeks)
Description: Participants will be assessed with the Generalized Anxiety Disorder 7 (GAD-7) at baseline, at 4 weeks, and at 8 weeks (posttreatment). (GAD-7 max-min scores=0-21, higher scores=worse outcome).
Time Frame: Baseline (T0), Weeks 3-4 (Midpoint, T1), Week 8 (Posttreatment, T2).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Score on the GAD-7
Arm/Group | Motherly App With Brief Psychotherapy | Educational App (Active Control)
Number analyzed (Participants) | 37 | 44
Score on the GAD-7
  T0 | 14.0 [12.8 to 15.3] | 13.5 [11.9 to 15.0]
  T1 | 11.1 [9.4 to 12.8] | 10.9 [9.3 to 12.6]
  T2 | 9.8 [7.8 to 11.8] | 9.7 [7.9 to 11.5]
Statistical Analysis 1: Comparison: Motherly App With Brief Psychotherapy vs Educational App (Active Control); Test type: Superiority; p = 0.910, t-test, 2 sided — Statistical tests were 2-sided and p values <0.05 were considered statistically significant; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Change in Maternal Prenatal Quality of Life From Baseline to Posttreatment (8 Weeks)
Description: Participants will be assessed with the 12-item health survey (SF-12) at baseline, at 4 weeks, and at 8 weeks (posttreatment). (SF-12 max-min scores=12-50, higher scores=worse outcome).
Time Frame: Baseline (T0), Weeks 3-4 (Midpoint, T1), Week 8 (Posttreatment, T2).
Population: This measure was not collected during all RCT due to logistics and the need to reduce data collection time.
Arm/Group | Motherly App With Brief Psychotherapy | Educational App (Active Control)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Maternal Prenatal Psychological Well-Being From Baseline to Posttreatment (8 Weeks).
Description: Participants were assessed with the Ryff's Psychological Well-Being Scale at baseline and at 8 weeks (posttreatment). (Ryff's Psychological Well-Being Scale max-min Total scores=36-216; higher scores=better outcome).
Time Frame: Baseline (T0), Week 8 (Posttreatment, T2).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Score on the PWB
Arm/Group | Motherly App With Brief Psychotherapy | Educational App (Active Control)
Number analyzed (Participants) | 37 | 44
Score on the PWB
  T0 | 149.7 [142.6 to 156.7] | 140.4 [133.1 to 147.7]
  T1 | 157.6 [149.7 to 165.4] | 153.0 [144.6 to 161.4]
Statistical Analysis 1: Comparison: Motherly App With Brief Psychotherapy vs Educational App (Active Control); Test type: Superiority; p = 0.442, t-test, 2 sided — Statistical tests were 2-sided and p values <0.05 were considered statistically significant; [statistical method as in outcome 1, analysis 1]

5. Secondary Outcome: Change in Maternal Physical Activity Levels From Baseline to Posttreatment (8 Weeks).
Description: Participants were assessed with the International Physical Activity Questionnaire (IPAQ) at baseline and at 8 weeks (posttreatment). (IPAQ measures Total Metabolic Equivalent of Task (MET) minutes per week (MET-min per week), higher MET-min per week=better outcome).
Time Frame: Baseline (T0), Week 8 (Posttreatment, T2).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: MET-min per week
Arm/Group | Motherly App With Brief Psychotherapy | Educational App (Active Control)
Number analyzed (Participants) | 37 | 44
MET-min per week
  T0 | 1626.0 [845.1 to 2407.0] | 2160.1 [1355.4 to 2964.8]
  T2 | 2770.0 [682.4 to 4859.0] | 1540.1 [1040.7 to 2039.5]
Statistical Analysis 1: Comparison: Motherly App With Brief Psychotherapy vs Educational App (Active Control); Test type: Superiority; p = 0.223, t-test, 2 sided — Statistical tests were 2-sided and p values <0.05 were considered statistically significant; [statistical method as in outcome 1, analysis 1]

6. Secondary Outcome: Change in Maternal Prenatal Perceived Stress From Baseline to Posttreatment (8 Weeks).
Description: Participants were assessed with the Perceived Stress Scale (PSS) at baseline, at 4 weeks, and at 8 weeks (posttreatment). (PSS max-min scores=0-40, higher scores=worse outcome).
Time Frame: Baseline (T0), Weeks 3-4 (Midpoint, T1), Week 8 (Posttreatment, T2).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Score on the PSS
Arm/Group | Motherly App With Brief Psychotherapy | Educational App (Active Control)
Number analyzed (Participants) | 37 | 44
Score on the PSS
  T0 | 26.5 [24.7 to 28.3] | 26.6 [24.6 to 28.6]
  T1 | 25.6 [23.5 to 27.7] | 25.0 [22.9 to 27.2]
  T2 | 23.9 [21.5 to 26.4] | 22.9 [20.6 to 25.2]
Statistical Analysis 1: Comparison: Motherly App With Brief Psychotherapy vs Educational App (Active Control); Test type: Superiority; p = 0.540, t-test, 2 sided — Statistical tests were 2-sided and p values <0.05 were considered statistically significant; [statistical method as in outcome 1, analysis 1]

7. Secondary Outcome: Change in Maternal Prenatal Depression Severity From Baseline to Posttreatment (8 Weeks).
Description: Participants were assessed with the Clinical Global Impressions Scale-Improvement (CGI-I). (scores in this scale are: 1=very much improved, 2= much improved, 3= minimally improved, 4 = no change, 5 = minimally worse, 6= much worse, 7= very much worse; scores were recoded as binary variable: improved (1, 2, 3) vs not-improved (4, 5, 6, 7).
Time Frame: Weeks 3-4 (Midpoint, T1), Week 8 (Posttreatment, T2).
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion (in percentage)
Arm/Group | Motherly App With Brief Psychotherapy | Educational App (Active Control)
Number analyzed (Participants) | 37 | 44
Proportion (in percentage)
  T1 | 63 [45 to 80] | 73 [59 to 87]
  T2 | 80 [65 to 94] | 80 [66 to 93]
Statistical Analysis 1: Comparison: Motherly App With Brief Psychotherapy vs Educational App (Active Control); Test type: Superiority; p = 0.901, t-test, 2 sided — Statistical tests were 2-sided and p values <0.05 were considered statistically significant; [statistical method as in outcome 1, analysis 1]

8. Secondary Outcome: Change in Maternal Prenatal Sleep Quality From Baseline to Posttreatment (8 Weeks).
Description: Participants were assessed with the Single-item Sleep Quality Scale (SIMP) at baseline, at 4 weeks, and at 8 weeks (posttreatment). (SIMP max-min scores=0-10, higher scores=better outcome).
Time Frame: Baseline (T0), Weeks 3-4 (Midpoint, T1), Week 8 (Posttreatment, T2).
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Score on SQA
Arm/Group | Motherly App With Brief Psychotherapy | Educational App (Active Control)
Number analyzed (Participants) | 37 | 44
Score on SQA
  T0 | 4.6 [4.0 to 5.2] | 4.6 [4.0 to 5.2]
  T1 | 5.6 [4.8 to 6.4] | 5.0 [4.3 to 5.8]
  T2 | 5.6 [4.7 to 6.5] | 5.4 [4.7 to 6.1]
Statistical Analysis 1: Comparison: Motherly App With Brief Psychotherapy vs Educational App (Active Control); Test type: Superiority; p = 0.748, t-test, 2 sided — Statistical tests were 2-sided and p values <0.05 were considered statistically significant; [statistical method as in outcome 1, analysis 1]

9. Secondary Outcome: Infant Developmental Milestones at 2 Months of Age.
Description: Child developmental milestones will be assessed with the Survey of Well-being of Young Children (SWYC) at 2 months of the child's age. (SWYC min-max=0-20, higher scores=better outcome).
Time Frame: When the infant is two months of age (Follow-up, T3).
Reporting Status: Not Posted

10. Secondary Outcome: Infant Social/Emotional Problems at 2 Months of Age.
Description: Infants will be assessed with the Baby Pediatric Symptom Checklist (BPSC) at 2 months of the child's age. (BPSC min-max=0-24, higher scores=worse outcome).
Time Frame: When the infant is two months of age (Follow-up, T3).
Reporting Status: Not Posted

11. Secondary Outcome: Change in Maternal Prenatal Depression From Baseline to Follow-up.
Description: Participants will be assessed with the Edinburgh Postnatal Depression Scale (EPDS) at baseline and when the infant is two months of age (Follow-up, T3). (EPDS max-min scores=0-30, higher scores=worse outcome).
Time Frame: Baseline (T0), when the infant is two months of age (Follow-up, T3).
Reporting Status: Not Posted

12. Secondary Outcome: Change in Maternal Prenatal Anxiety From Baseline to to Follow-up.
Description: Participants will be assessed with the Generalized Anxiety Disorder 7 (GAD-7) at baseline and when the infant is two months of age (Follow-up, T3). (GAD-7 max-min scores=0-21, higher scores=worse outcome).
Time Frame: Baseline (T0), when the infant is two months of age (Follow-up, T3).
Reporting Status: Not Posted

13. Secondary Outcome: Change in Maternal Prenatal Quality of Life From Baseline to to Follow-up.
Description: Participants will be assessed with the 12-item health survey (SF-12) at baseline and when the infant is two months of age (Follow-up, T3). (SF-12 max-min scores=12-50, higher scores=worse outcome).
Time Frame: Baseline (T0), when the infant is two months of age (Follow-up, T3).
Reporting Status: Not Posted

14. Secondary Outcome: Change in Maternal Prenatal Psychological Well-Being From Baseline to Follow-up.
Description: Participants will be assessed with the Ryff's Psychological Well-Being Scale at baseline and when the infant is two months of age (Follow-up, T3). (Ryff's Psychological Well-Being Scale max-min scores=6-36, higher scores=better outcome).
Time Frame: Baseline (T0), when the infant is two months of age (Follow-up, T3).
Reporting Status: Not Posted

15. Secondary Outcome: Change in Maternal Prenatal Perceived Stress From Baseline to Follow-up.
Description: Participants will be assessed with the Perceived Stress Scale (PSS) at baseline and when the infant is two months of age (Follow-up, T3). (PSS max-min scores=0-40, higher scores=worse outcome).
Time Frame: Baseline (T0), when the infant is two months of age (Follow-up, T3).
Reporting Status: Not Posted

16. Secondary Outcome: Change in Maternal Prenatal Depression Severity From Baseline to Follow-up.
Description: Participants will be assessed with the Clinical Global Impressions Scale-Improvement (CGI-I) when the infant is two months of age (Follow-up, T3). (CGI-I, min-max=0-7, higher scores=worst outcome).
Time Frame: Baseline (T0), when the infant is two months of age (Follow-up, T3).
Reporting Status: Not Posted

17. Secondary Outcome: Change in Maternal Prenatal Sleep Quality From Baseline to Follow-up.
Description: Participants will be assessed with the Single-item Sleep Quality Scale (SIMP) at baseline and when the infant is two months of age (Follow-up, T3). (SIMP max-min scores=0-10, higher scores=better outcome).
Time Frame: Baseline (T0), when the infant is two months of age (Follow-up, T3).
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the trial by psychotherapist during their sessions with participants. Moreover, assessors collected information on adverse events during the assessments at baseline (T0), mid-treatment (T1), posttreatment (T3).
Description: Given that the intervention in this study is non-invasive, with a very low risk for participants of serious adverse events and mortality, then adverse events were collected qualitatively throughout the trial by the assessors, who asked participants about psychological distress and discomfort from the interventions.
Arm/Group | Motherly App With Brief Psychotherapy | Educational App (Active Control)
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/44
Other Adverse Events (participants affected / at risk) | 0/37 | 0/44

LIMITATIONS AND CAVEATS:
sample was primarily composed of highly educated women with high family income. Therefore, considering Brazil is a LMIC with inequality and widespread poverty, it is difficult to generalize our findings to other regions and countries. Study was conducted during the COVID-19 pandemic, which may have impacted participants' mental health.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-07-31): https://cdn.clinicaltrials.gov/large-docs/66/NCT04495166/Prot_SAP_ICF_000.pdf